CLINICAL TRIAL: NCT02266043
Title: Cohort Study on Prevalence and Early Treatment Outcomes in Pierre-Robin-Like Phenotype
Brief Title: Early Treatment Outcomes in Pierre-Robin-Like Phenotype
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: FACE-Subproject SP5-Tuebingen
Record Dates: First submitted 2014-09-30; First posted 2014-10-16 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Pierre Robin Syndrome
Keywords: Upper airway obstruction
MeSH Terms: conditions — Pierre Robin Syndrome; Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pre-epiglottic baton plate (PEBP) — modified acrylic palatal plate in which a velar extension resembling a spur or baton shifts the base of the tongue forward.
  This treatment is the standard care for infants with Pierre-Robin-Like Phenotype in the participating study centers and not assigned by protocol.

SUMMARY:
In a longitudinal cohort study, we want to assess the effect of the pre-epiglottic baton plate, the main treatment approach currently used in Germany for Pierre-Robin-Like phenotype, on upper airway obstruction and failure to thrive using objective criteria (mixed-obstructive apnea index assessed by polysomnography, standard deviation score for body weight) upon admission and 3 months after hospital discharge.

DETAILED DESCRIPTION:
Pierre-Robin sequence consists of a small lower jaw, a retropositioned tongue (glossoptosis), and optionally cleft palate, leading to severe upper airway obstruction and failure to thrive; occasionally even to sudden infant death. Treatment approaches are heterogeneous, some are considerably invasive; few have been evaluated by objective tests.

In a longitudinal cohort study, we want to assess the effect of the pre-epiglottic baton plate on upper airway obstruction and failure to thrive using objective criteria (mixed-obstructive apnea index assessed by polysomnography, standard deviation score for body weight) upon admission and 3 months after hospital discharge. The pre-epiglottic baton plate is the main treatment approach currently used in Germany for this condition and practised standard care in the three participating study centers.

These data will help to compare the effect of the main treatment currently used in Germany with international data on more invasive treatments used in this rare condition.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 1 year at admission, Pierre-Robin-like phenotype

Exclusion Criteria:

* no parental consent; need for immediate tracheotomy

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants <1 year admitted with Pierre-Robin-like phenotype to participating centres
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in mixed-obstructive apnea index (MOAI) | upon admission within the first year of life (before start of treatment) and 3 months after hospital discharge
  Change in mixed-obstructive apnea index (MOAI) assessed by polygraphy from pre- to post-intervention as a marker of Pierre-Robin-sequence-related breathing disorder

SECONDARY OUTCOMES:
Change in standard deviation score for body weight | upon admission within the first year of life (before start of treatment) and 3 months after hospital discharge
  Body weight will be obtained by electronic scales and the standard deviation score for weight calculated
Duration of hospital stay | admission within the first year of life for initiation of study intervention
Treatment failure | 3 months after admission for initiation of study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christian F Poets, MD, Principal Investigator — Dept. of Neonatology and Interdisciplinary Centre forCraniofacial Malformations, University Hospital Tuebingen; Siegmar Reinert, MD, PhD, Principal Investigator — Dept. of Craniofacial Surgery, University Hospital Tuebingen
Locations (3):
- Germany (3):
  - Centre of Competence for Oro- and Craniofacial Malformations and Department of Neonatology, Univ. Hospital of Cologne, Cologne
  - Dept. of Neonatology and Interdisciplinary Centre for Craniofacial Malformations, University Hospital Tuebingen, Tübingen
  - Dept. of Orthodontics and University Children's Hospital, University Hospital of Wuerzburg, Würzburg

REFERENCES:
- [Derived] Poets CF, Maas C, Buchenau W, Arand J, Vierzig A, Braumann B, Muller-Hagedorn S. Multicenter study on the effectiveness of the pre-epiglottic baton plate for airway obstruction and feeding problems in Robin sequence. Orphanet J Rare Dis. 2017 Mar 9;12(1):46. doi: 10.1186/s13023-017-0602-8. PMID 28274235